CLINICAL TRIAL: NCT03432221
Title: Efficacy Of Switching From SSRI to Desvenlafaxine on Cognitive Function In Patients With an Acute Episode of Major Depression
Brief Title: Switching From SSRI to Desvenlafaxine on Cognitive Functioning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Narcis Cardoner, MD, PhD, Narcís Cardoner, MD, PhD, Corporacion Parc Tauli
Other Study IDs: 2017.116
Record Dates: First submitted 2018-01-08; First posted 2018-02-14 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Major Depressive Disorder
Keywords: Cognition, antidepressants drugs, SNRI, hot cognition, functioning
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MDD: Patients who met DSM-5 criteria for MDD attending the outpatient psychiatric service of the Hospital Universitari Parc Taulí. Patients must have a lack of response to SSRI (Maximize dose for adequate time), being the next therapeutic option the introduction of desvenlafaxine.
  Interventions: Drug: Desvenlafaxine
- Healthy Controls: Healthy participants matched by age, gender and educational level without history of psychiatric disorders and no familial history of mood disorders will be recruited

INTERVENTIONS:
Drug: Desvenlafaxine — Patients included in the study will receive antidepressant treatment with desvenlafaxine. The switch from SSRI to desvenlafaxine will coincide with the baseline visit (Visit 0). The dose of desvenlafaxine will be established based on clinical judgment. As the approach will be naturalistic, the inclusion in this study will not influence the clinical choice, hence changes in the pharmacological strategy will be permitted.
  Groups: MDD

SUMMARY:
Given the importance of cognitive function on depressed patients' treatment outcome and return to premorbid functioning, the effect of antidepressant drugs on cognition has become of primary concern. The aim of the present study is to assess the clinical outcome of switching from a selective serotonin reuptake inhibitor (SSRI) to desvenlafaxine on cognitive function in a Spanish sample of adults with moderate to severe major depressive disorder (MDD).

This open-label clinical study will include a total of 36 MDD outpatients receiving treatment with desvenlafaxine according to treating psychiatrist clinical judgment.

The primary efficacy endpoint will be changes from baseline to week 12 in cognitive function measured by a composite z-score comprising the Digit Symbol Substitution Test (DSST) and Rey Auditory Verbal Learning Test (RAVLT) scores. The secondary efficacy endpoints will involve depression severity, additional measures of subjective and objective cognitive function (including cold and hot cognitive function tasks), and functional status.

A matched sample of 36 healthy controls will be assessed in order to obtain reference data for all cognitive function measurements. Patients with MDD and healthy controls will be compared regarding cognitive function both at baseline and after 12 weeks.

DETAILED DESCRIPTION:
BACKGROUND

Depression is a significant contributor to the global burden of disease and affects people in all communities across the world. Today, depression is estimated to affect 350 million people. The World Mental Health Survey conducted in 17 countries found that, on average, about 1 in 20 people reported having an episode of depression in the previous year. Depressive disorders often start at a young age; drastically reduce people's functioning and often are recurring. For all these reasons, depression is the leading cause of disability worldwide in terms of total years lost due to disability.

Commonly the diagnosis and treatment of major depressive disorder is based on mood symptoms. However, cognitive impairments are often present in this disorder. In this respect, the recent Diagnostic and Statistical Manual 5 (DSM-5) highlight impairment in cognitive function as a criterion in the diagnosis of a major depressive episode (MDE) (American Psychiatric Association. At clinical level, patients frequently present subjective complaints during and after resolution of an MDE. Moreover, objective deficits measured by neuropsychological tests are also reported in different cognitive domains in cold cognitive function - executive function, processing speed, attention, learning or memory- (Hammar &Ardal, 2009) or also in hot cognitive function -negative biases in perception, attention and memory, and aberrant reward/punishment processing-.

Different meta-analyses have demonstrated that these deficits may emerge from the first depressive episode with relevant intensification during each acute MDE persisting in some depressive patients even during the resolution of the acute episode. These deficits, both in an acute episode and in remission, have a relevant impact on clinical and functional outcomes, in the first case by reducing the chance to fully recover and in the second by increasing the risk of relapse. Moreover, cognitive deficits have shown to have a negative influence in functional performance in academic, social and working life (Lee et al., 2013,). In this context, recent studies have shown that a larger number of MDD episodes, a longer duration of illness and a poor response to antidepressant treatments might explain the maintenance of cognitive dysfunction, even in patients with some clinical response.

Persistent cognitive deficits in depression play a crucial role in some patients׳ ability to achieve a functional recovery. With this respect, cognitive function in depression is significantly also related to employment status. A preliminary study suggests that deficits in executive functioning have a mediating effect on the relationship between depression and impaired activities of daily living. Moreover, mood disorder patients with neuropsychological deficits tend to be less compliant with antidepressant treatment (Martinez-Aran et al., 2009) and show an increased risk for suicide. In this context, the identification and treatment of specific cognitive deficits may be a cardinal aspect in the achievement of depression recovery and, even more important, in the functional normalization of patients to their pre-morbid levels.

At present there is a growing interest on the role of antidepressant treatment in the modulation of cognitive deficits associated with depression. Despite the wide array of effective antidepressant agents, the knowledge on the impact of available drugs on cognitive function constitutes a relevant unmet need. Indeed, the number of studies focusing on this issue is relatively scarce and the outcome of cognitive symptoms is widely variable. Potential pro-cognitive effect of a particular antidepressant mostly relay on its specific mechanisms of action, anf in the last years the evidence accumulated have support that drug involving more targets such as dual (duloxetine) or multimodal (vortioxetine) antidepressants show more pro-cognitive properties than those with one major mechanism (SSRI).

However, the clinical studies putting cognitive dysfunction as the primary outcome in depression trials are scarce and further support of these initial promising findings of the effects of dual/multimodal antidepressants on cognition are required.

OBJECTIVES

This open-label clinical study will evaluate the clinical outcome of switching to desvenlafaxine on cognitive function of patients with major depressive disorder with inadequate response to selective serotonin reuptake inhibitor (SSRI)

* Primary Objective

To study differences in cognitive function in moderate to severe MDD patients with inadequate response to SSRI and healthy controls at baseline and after 12 weeks of treatment with desvenlafaxine.

* Secondary Objective

To study differences in subjective cognitive function (cognitive complains), measured by PDQ-5 at baseline and after 12 weeks of treatment with Desvenlafaxine.

To study differences in cognitive function, measured by neuropsychological tests battery (including cold and hot cognitive function) at baseline and after 12 weeks of treatment with desvenlafaxine.

To study differences in depression severity, measured HDRS-17 and CGI at baseline and after 12 weeks of treatment with desvenlafaxine.

To study changes in subjective remission and functional status measured with Remission Depression Questionnaire (RDQ) and the Short Assessement Functioning Test (FAST), respectively.

ELIGIBILITY:
Inclusion Criteria:

1. MDD Patients in whom switching to desvenlafaxine is considered by treating psychiatrist as the next treatment option.
2. MDD diagnostic confirmation with the mini-international neuropsychiatric interview (MINI) (Sheehan et al., 1998),
3. Age range between 18 and 60
4. Non-response or incomplete response to a treatment with an SSRI in the current episode.
5. Score of 18 points or higher in the Hamilton depression rating scale (HAM-D-17) (Hamilton, 1967).

Exclusion Criteria:

1. Subjects will be excluded if they met criteria or had past history for the following disorders: posttraumatic stress disorder, obsessive-compulsive disorder, schizophrenia, psychotic, delusional, bipolar or substance abuse disorders. MINI will be used to exclude these potentially comorbid disorders.
2. Subjects with any present or past disease involving the nervous central system
3. A clinically significant unstable illness or clinically significant abnormal vital signs as determined by the investigator
4. Women entering the study could not be pregnant, and had to be oral contraceptive-free.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients attending at the outpatient unit at the Psychiatry Department of the Hospital Universitari Parc Taulí will be consecutively recruited until the study sample (36) is reached.
  Healthy controls will be seek from the same socio-demographic environment as patients (Vallès area, Spain)
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-06-03 (Estimated); Study Completion 2019-06-03 (Estimated)

PRIMARY OUTCOMES:
Composite cognitive measure | Change from baseline to 12 weeks
  Composite z-score (Digit Symbol Substitution Test (DSST) + Rey Auditory Verbal Learning Test (RAVLT))

SECONDARY OUTCOMES:
Subjective cognitive function | Baseline, 2nd week, 4th week, 6th week, 8th week, 10th week, 12th week
  Perceived deficit Questionnaire short version (PDQ-5)
Attention | Baseline and after 12 weeks
  Attention (Digits subtest forward -WAIS-IV- + Trail Making Test-A, TMT-A)
Processing speed | Baseline and after 12 weeks
  Psychomotor velocity (Digit Symbol Substitution Test, DSST)
Verbal Memory | Baseline and after 12 weeks
  Memory cognitive domain explored with:
  - Rey Auditory Verbal Learning Test (Verbal)
Executive Functions | Baseline and after 12 weeks
  Composite score composed by: Trail Making Test-B + Phonetic fluency & semantic fluency + Wisconsin Card Sorting Test
Hot cognition | Baseline and after 12 weeks
  Emotion recognition ability explored with:
  - Pictures of Facial Affect (POFA)
Intelligence quotient | Baseline
  Measure of pre-morbid intelligence (Vocabulary (WAIS IV) + Block Design (WAIS-IV))
Depressive symptoms | Baseline, 2nd week, 4th week, 6th week, 8th week, 10th week, 12th week
  The Hamilton Depression Rating Scale, 17 items (HDRS), designed to rate the severity of depression in patients.
  0 - 7 = Normal 8 - 13 = Mild Depression 14-18 = Moderate Depression 19 - 22 = Severe Depression >23 = Very Severe Depression
Anxiety symptoms | Baseline, 2nd week, 4th week, 6th week, 8th week, 10th week, 12th week
  The Hamilton Anxiety Rating Scale (HAM-A), to measure the severity of anxiety symptoms.
  14-17 = Mild Anxiety 18-24 = Moderate Anxiety 25-30 = Severe Anxiety
Severity and improvement of depression | Baseline, 2nd week, 4th week, 6th week, 8th week, 10th week, 12th week
  The Clinical Global Impression (CGI)
Self-perceived remission status | Baseline, 2nd week, 4th week, 6th week, 8th week, 10th week, 12th week
  The Remission from Depression Questionnaire (RDQ)
Disability | Baseline and after 12 weeks
  Functional disability measured with the Sheehan Disability Scale (SDS) SDS: developed to assess functional impairment in three inter-related domains; work/school, social and family life. The 3 items can also be summed into a single dimensional measure of global functional impairment that rages from 0 (unimpaired) to 30 (highly impaired).
Functioning | Baseline and after 12 weeks
  Functioning Assessment Short Test (FAST)
  FAST: brief instrument designed to assess the main functioning problems experienced by psychiatric patients, particularly those with mood disorders. Scores > 11(out of 75)= Impairment.
Sexual dysfunction | Baseline and after 12 weeks
  The Arizona Sexual Experience Scale (ASEX): a five-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm.
Side effect rating scale for psychotropic drugs | Baseline, 2nd week, 4th week, 6th week, 8th week, 10th week, 12th week
  The UKU side effect rating scale: A Comprehensive Rating Scale for Psychotropic Drugs and a Cross-sectional Study of Side Effects in Neuroleptic-treated Patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Corporació Sanitària Parc Taulí, Sabadell, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baune BT, Miller R, McAfoose J, Johnson M, Quirk F, Mitchell D. The role of cognitive impairment in general functioning in major depression. Psychiatry Res. 2010 Apr 30;176(2-3):183-9. doi: 10.1016/j.psychres.2008.12.001. PMID 20138370
- [Background] Bora E, Harrison BJ, Yucel M, Pantelis C. Cognitive impairment in euthymic major depressive disorder: a meta-analysis. Psychol Med. 2013 Oct;43(10):2017-26. doi: 10.1017/S0033291712002085. Epub 2012 Oct 26. PMID 23098294
- [Background] Ferguson JM, Wesnes KA, Schwartz GE. Reboxetine versus paroxetine versus placebo: effects on cognitive functioning in depressed patients. Int Clin Psychopharmacol. 2003 Jan;18(1):9-14. doi: 10.1097/00004850-200301000-00002. PMID 12490769
- [Background] Hammar A, Ardal G. Cognitive functioning in major depression--a summary. Front Hum Neurosci. 2009 Sep 25;3:26. doi: 10.3389/neuro.09.026.2009. eCollection 2009. PMID 19826496
- [Background] Herrera-Guzman I, Gudayol-Ferre E, Herrera-Abarca JE, Herrera-Guzman D, Montelongo-Pedraza P, Padros Blazquez F, Pero-Cebollero M, Guardia-Olmos J. Major Depressive Disorder in recovery and neuropsychological functioning: effects of selective serotonin reuptake inhibitor and dual inhibitor depression treatments on residual cognitive deficits in patients with Major Depressive Disorder in recovery. J Affect Disord. 2010 Jun;123(1-3):341-50. doi: 10.1016/j.jad.2009.10.009. Epub 2009 Nov 6. PMID 19896719
- [Background] Herrera-Guzman I, Gudayol-Ferre E, Herrera-Guzman D, Guardia-Olmos J, Hinojosa-Calvo E, Herrera-Abarca JE. Effects of selective serotonin reuptake and dual serotonergic-noradrenergic reuptake treatments on memory and mental processing speed in patients with major depressive disorder. J Psychiatr Res. 2009 Jun;43(9):855-63. doi: 10.1016/j.jpsychires.2008.10.015. Epub 2009 Jan 6. PMID 19128810
- [Background] Jaeger J, Berns S, Uzelac S, Davis-Conway S. Neurocognitive deficits and disability in major depressive disorder. Psychiatry Res. 2006 Nov 29;145(1):39-48. doi: 10.1016/j.psychres.2005.11.011. Epub 2006 Oct 11. PMID 17045658
- [Background] Kiosses DN, Alexopoulos GS. IADL functions, cognitive deficits, and severity of depression: a preliminary study. Am J Geriatr Psychiatry. 2005 Mar;13(3):244-9. doi: 10.1176/appi.ajgp.13.3.244. PMID 15728756
- [Background] Lee RS, Hermens DF, Porter MA, Redoblado-Hodge MA. A meta-analysis of cognitive deficits in first-episode Major Depressive Disorder. J Affect Disord. 2012 Oct;140(2):113-24. doi: 10.1016/j.jad.2011.10.023. Epub 2011 Nov 15. PMID 22088608
- [Background] Levkovitz Y, Caftori R, Avital A, Richter-Levin G. The SSRIs drug Fluoxetine, but not the noradrenergic tricyclic drug Desipramine, improves memory performance during acute major depression. Brain Res Bull. 2002 Aug 15;58(4):345-50. doi: 10.1016/s0361-9230(01)00780-8. PMID 12183009
- [Background] Martinez-Aran A, Scott J, Colom F, Torrent C, Tabares-Seisdedos R, Daban C, Leboyer M, Henry C, Goodwin GM, Gonzalez-Pinto A, Cruz N, Sanchez-Moreno J, Vieta E. Treatment nonadherence and neurocognitive impairment in bipolar disorder. J Clin Psychiatry. 2009 Jul;70(7):1017-23. doi: 10.4088/JCP.08m04408. Epub 2009 Jun 2. PMID 19497247
- [Background] McIntyre RS, Lophaven S, Olsen CK. A randomized, double-blind, placebo-controlled study of vortioxetine on cognitive function in depressed adults. Int J Neuropsychopharmacol. 2014 Oct;17(10):1557-67. doi: 10.1017/S1461145714000546. Epub 2014 Apr 30. PMID 24787143
- [Background] Miskowiak KW, Carvalho AF. 'Hot' cognition in major depressive disorder: a systematic review. CNS Neurol Disord Drug Targets. 2014;13(10):1787-803. doi: 10.2174/1871527313666141130205713. PMID 25470389
- [Background] Nierenberg AA, Husain MM, Trivedi MH, Fava M, Warden D, Wisniewski SR, Miyahara S, Rush AJ. Residual symptoms after remission of major depressive disorder with citalopram and risk of relapse: a STAR*D report. Psychol Med. 2010 Jan;40(1):41-50. doi: 10.1017/S0033291709006011. Epub 2009 May 22. PMID 19460188
- [Background] Roiser JP, Sahakian BJ. Hot and cold cognition in depression. CNS Spectr. 2013 Jun;18(3):139-49. doi: 10.1017/S1092852913000072. Epub 2013 Mar 12. PMID 23481353
- [Background] Trivedi MH, Greer TL. Cognitive dysfunction in unipolar depression: implications for treatment. J Affect Disord. 2014 Jan;152-154:19-27. doi: 10.1016/j.jad.2013.09.012. Epub 2013 Sep 25. PMID 24215896
- [Background] Wagner S, Doering B, Helmreich I, Lieb K, Tadic A. A meta-analysis of executive dysfunctions in unipolar major depressive disorder without psychotic symptoms and their changes during antidepressant treatment. Acta Psychiatr Scand. 2012 Apr;125(4):281-92. doi: 10.1111/j.1600-0447.2011.01762.x. Epub 2011 Oct 18. PMID 22007857
- [Background] Westheide J, Quednow BB, Kuhn KU, Hoppe C, Cooper-Mahkorn D, Hawellek B, Eichler P, Maier W, Wagner M. Executive performance of depressed suicide attempters: the role of suicidal ideation. Eur Arch Psychiatry Clin Neurosci. 2008 Oct;258(7):414-21. doi: 10.1007/s00406-008-0811-1. Epub 2008 Mar 11. PMID 18330667
- [Derived] Vicent-Gil M, Trujols J, Sagues T, Serra-Blasco M, Navarra-Ventura G, Mantellini CL, Crivilles S, Portella MJ, Cardoner N. Insights on the cognitive enhancement effect of desvenlafaxine in major depressive disorder. Ann Gen Psychiatry. 2025 Mar 19;24(1):16. doi: 10.1186/s12991-025-00552-2. PMID 40108685